CLINICAL TRIAL: NCT04948697
Title: A Phase 2, Randomized, Open-labeled Clinical Study Investigating the Efficacy and Safety of Ociperlimab in Combination With Tislelizumab Plus BAT1706 and of Tislelizumab Plus BAT1706 as First-line Treatment in Patients With Advanced Hepatocellular Carcinoma
Brief Title: A Study Investigating the Efficacy and Safety of Ociperlimab and Tislelizumab and BAT1706 Combinations in Patients With Advanced HCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AdvanTIG-206; CTR20211546 (Registry Identifier: ChinaDrugTrials)
Record Dates: First submitted 2021-06-20; First posted 2021-07-02 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-01

CONDITIONS: Advanced Hepatocellular Carcinoma
MeSH Terms: interventions — tislelizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Ociperlimab + Tislelizumab + BAT1706 (Experimental): Participants received tislelizumab 200 milligrams (mg) intravenously once every 3 weeks followed by BAT1706 15 milligrams per kilogram (mg/kg) intravenously once every 3 weeks followed by ociperlimab 900 mg intravenously once every 3 weeks in 21-day treatment cycles until disease progression, unacceptable toxicity, or withdrawal for other reasons, whichever occurred first.
  Interventions: Drug: Ociperlimab; Drug: Tislelizumab; Drug: BAT1706
- Arm B: Tislelizumab + BAT1706 (Experimental): Participants received tislelizumab 200 mg intravenously once every 3 weeks followed by BAT1706 15 mg/kg intravenously once every 3 weeks in 21-day treatment cycles until disease progression, unacceptable toxicity, or withdrawal for other reasons, whichever occurred first.
  Interventions: Drug: Tislelizumab; Drug: BAT1706

INTERVENTIONS:
Drug: Ociperlimab — 900 mg intravenously once every 3 weeks (dosed in 21-day cycles)
  Other Names: BGB-A1217
  Arms: Arm A: Ociperlimab + Tislelizumab + BAT1706
Drug: Tislelizumab — 200 mg intravenously once every 3 weeks (dosed in 21-day cycles)
  Other Names: BGB-A317
Drug: BAT1706 — 15 mg/kg intravenously once every 3 weeks (dosed in 21-day cycles)
  Other Names: Bevacizumab Injection

SUMMARY:
This was a Phase 2, randomized, multicenter, open-label, 2-arm study to investigate the efficacy and safety of ociperlimab in combination with tislelizumab plus BAT1706, and tislelizumab plus BAT1706, as first-line treatment in participants with advanced Hepatocellular Carcinoma (HCC).

ELIGIBILITY:
Criteria:

Inclusion Criteria:

1. Histologically confirmed HCC
2. Barcelona Clinic Liver Cancer (BCLC) Stage C disease, or BCLC Stage B disease that was not amenable to or had progressed after loco-regional therapy, and was not amenable to a curative treatment approach
3. Tumor tissue required for an evaluable programmed cell death protein-ligand 1 (PD-L1) expression result
4. No prior systemic therapy for HCC
5. At least 1 measurable lesion as defined per RECIST v1.1
6. Adequate organ function during screening and before randomization

Exclusion Criteria:

1. Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC histology
2. Prior therapy with antibody or drug specifically targeting T-cell costimulation or checkpoint pathway; prior treatment with bevacizumab or its biosimilars
3. Prior history of >= Grade 2 hepatic encephalopathy
4. Leptomeningeal disease or uncontrolled, untreated brain metastasis
5. Active autoimmune diseases or history of autoimmune diseases that may relapse
6. History of interstitial lung disease, non-infectious pneumonitis or uncontrolled lung diseases including pulmonary fibrosis, acute lung diseases
7. Infection (including tuberculosis) requiring systemic antibacterial, antifungal, or antiviral therapy within 14 days of randomization
8. Prior allogeneic stem cell transplantation or organ transplantation
9. Significant cardiovascular risk factors
10. Untreated or incompletely treated esophageal or gastric varices with bleeding or high risk of bleeding
11. History of severe hypersensitivity reactions to other monoclonal antibodies
12. Administered a live vaccine <=28 days before randomization

NOTE: Other protocol Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (28):
- China (23):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chongqing Three Gorges Central Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Mengchao Hepatobiliary Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First Affiliated Hospital, Sun Yat Sen University, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Affiliated Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Tianjin Third Central Hospital, Tianjin, Tianjin Municipality
  - Karamay Central Hospital of Xinjiang, Karamay, Xinjiang
  - Zhejiang University College of Medicine Second Affiliated Hospital, Hangzhou, Zhejiang
  - Zhejiang Provincial Peoples Hospital, Hangzhou, Zhejiang
  - Huzhou Central Hospital, Huzhou, Zhejiang
  - Jinhua Municipal Central Hospital, Jinhua, Zhejiang
  - Hwa Mei Hospital, University of Chinese Academy of Sciences (Ningbo No Hospital), Ningbo, Zhejiang
- Taiwan (5):
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Medical Center, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 94 eligible participants were randomized in a 2:1 ratio to receive ociperlimab in combination with tislelizumab + BAT1706 or tislelizumab + BAT1706.
Pre-assignment Details: Randomization was stratified according to programmed cell death protein-ligand 1 (PD-L1) expression and macrovascular invasion (MVI)/extrahepatic spread (EHS) (present versus absent) status.
Period: Overall Study
Arm/Group | Arm A: Ociperlimab + Tislelizumab + BAT1706 | Arm B: Tislelizumab + BAT1706
Started | 62 | 32
Treated | 62 | 31
Completed | 0 | 0
Not Completed | 62 | 32
Not completed — Progressive disease | 27 | 18
Not completed — Adverse Event | 14 | 4
Not completed — Participant moved to long term extension study | 7 | 4
Not completed — Withdrawal by Subject | 10 | 0
Not completed — Closed by Sponsor | 3 | 2
Not completed — Physician Decision | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Other-Miscellaneous | 1 | 0
Not completed — Randomized but not treated | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on Intent-to-Treat (ITT) analysis set that included all randomized participants and were analyzed according to their randomized treatment arm (i.e., Arm A or Arm B).
Groups:
- Arm A: Ociperlimab + Tislelizumab + BAT1706: Participants received tislelizumab 200 mg intravenously once every 3 weeks followed by BAT1706 15 mg/kg intravenously once every 3 weeks followed by ociperlimab 900 mg intravenously once every 3 weeks in 21-day treatment cycles until disease progression, unacceptable toxicity, or withdrawal for other reasons, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | Arm A: Ociperlimab + Tislelizumab + BAT1706 | Arm B: Tislelizumab + BAT1706 | Total
Number analyzed (Participants) | 62 | 32 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (11.27) | 59.1 (10.77) | 58.6 (11.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 57 | 30 | 87
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 62 | 32 | 94
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 62 | 32 | 94
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Macrovascular invasion (MVI) Status [Count of Participants; unit: Participants]
  Present | 13 | 12 | 25
  Absent | 49 | 20 | 69
Extrahepatic spread (EHS) Status [Count of Participants; unit: Participants]
  Present | 31 | 19 | 50
  Absent | 31 | 13 | 44

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) as Assessed by the Investigator
Description: ORR was defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) per response evaluation criteria in solid tumors version(v) 1.1 (RECIST v1.1). Per RECIST v1.1., CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 millimeters (mm). PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first (i.e., up to 27 months)
Population: Analysis was performed on the Intent-to-Treat (ITT) analysis set that included all randomized participants and were analyzed according to their randomized treatment arm (i.e., Arm A or Arm B).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Ociperlimab + Tislelizumab + BAT1706 | Arm B: Tislelizumab + BAT1706
Number analyzed (Participants) | 62 | 32
percentage of participants | 37.1 [25.2 to 50.3] | 40.6 [23.7 to 59.4]

2. Secondary Outcome: Duration Of Response (DOR) as Assessed by the Investigator
Description: DOR was defined as the time from the date of first documentation of a partial response (PR) or better to the date of first documentation of progressive disease or death whichever comes first, assessed based on RECIST v1.1. Median DOR was estimated using the Kaplan-Meier method. Per RECIST v1.1, PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Progressive disease was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study.
Time Frame: From the first confirmed objective response until the first documentation of disease progression or death, whichever came first (i.e. up to 27 months)
Population: Analysis was performed on participants in the ITT analysis set with an objective response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Ociperlimab + Tislelizumab + BAT1706 | Arm B: Tislelizumab + BAT1706
Number analyzed (Participants) | 23 | 13
months | 12.6 [6.9 to NA] — Upper limit of 95% confidence interval (CI) could not be estimated due to low number of participants with an event. | 12.4 [5.4 to NA] — Upper limit of 95% CI could not be estimated due to low number of participants with an event.

3. Secondary Outcome: Time to Response (TTR) as Assessed by the Investigator
Description: TTR was defined as the time from the randomization date to the date of first documented partial response (PR) or better by the investigator, assessed based on RECIST v1.1. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the randomization date to the first documentation of response (up to 27 months)
Population: Analysis was performed on participants in the ITT analysis set with an objective response.
Measure: Median (Full Range); unit: months
Arm/Group | Arm A: Ociperlimab + Tislelizumab + BAT1706 | Arm B: Tislelizumab + BAT1706
Number analyzed (Participants) | 23 | 13
months | 2.76 [1.2 to 6.9] | 4.17 [1.4 to 8.3]

4. Secondary Outcome: Disease Control Rate (DCR) as Assessed by the Investigator
Description: DCR was defined as the percentage of participants who achieve complete response (CR), partial response (PR) or stable disease (SD), assessed based on RECIST v1.1. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: as for outcome 1
Population: Analysis was performed on ITT analysis set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Ociperlimab + Tislelizumab + BAT1706 | Arm B: Tislelizumab + BAT1706
Number analyzed (Participants) | 62 | 32
percentage of participants | 77.4 [65.0 to 87.1] | 71.9 [53.3 to 86.3]

5. Secondary Outcome: Clinical Benefit Rate (CBR) as Assessed by the Investigator
Description: CBR was defined as the percentage of participants who achieve complete response (CR), partial response (PR), or durable stable disease (stable disease defined as >= 24 weeks). Per RECIST 1.1., CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: as for outcome 1
Population: Analysis was performed on ITT analysis set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Ociperlimab + Tislelizumab + BAT1706 | Arm B: Tislelizumab + BAT1706
Number analyzed (Participants) | 62 | 32
percentage of participants | 59.7 [46.4 to 71.9] | 56.3 [37.7 to 73.6]

6. Secondary Outcome: Progression-Free Survival (PFS) as Assessed by the Investigator
Description: PFS was evaluated by the investigator according to RECIST version 1.1; and was defined as the time from the randomization date to the date of first documentation of disease progression or date of death from any cause, whichever occurred first. Median PFS was estimated using the Kaplan-Meier method. Per RECIST v 1.1, progressive disease was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study.
Time Frame: From the randomization date to the date of first documentation of disease progression or death, whichever came first (i.e., up to 27 months)
Population: Analysis was performed on ITT analysis set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Ociperlimab + Tislelizumab + BAT1706 | Arm B: Tislelizumab + BAT1706
Number analyzed (Participants) | 62 | 32
months | 8.3 [5.5 to 10.3] | 6.9 [4.1 to 17.4]

7. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the randomization date until the date of death from any cause. Median OS was estimated using the Kaplan-Meier method.
Time Frame: From the randomization date until the date of death from any cause (up to 27 months)
Population: Analysis was performed on ITT analysis set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Ociperlimab + Tislelizumab + BAT1706 | Arm B: Tislelizumab + BAT1706
Number analyzed (Participants) | 62 | 32
months | 19.7 [18.4 to NA] — Upper limit of 95% CI was not calculated due to low number of participants with events. | 22.9 [14.4 to NA] — Upper limit of 95% CI was not calculated due to low number of participants with events.

8. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: A TEAE was defined as an adverse event (AE) that had an onset date or a worsening in severity from baseline (pretreatment) on or after the first dose of study drug(s) and up to 30 days after the last dose of study drug(s), or initiation of new anticancer therapy, whichever occurs first. AEs were graded for severity using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version (v) 5.0, where Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4 - Life-threatening consequences; and Grade 5: Death related to AE. The TEAEs leading to death in this data table exclude death due to disease under study.
Time Frame: From the date of the first dose of study drug up to 30 days after last dose of study drug (i.e., up to 27 months)
Population: Analysis was performed on safety analysis set that included all participants of each arm who received at least 1 dose of study drugs.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Ociperlimab + Tislelizumab + BAT1706 | Arm B: Tislelizumab + BAT1706
Number analyzed (Participants) | 62 | 31
Participants
  TEAEs | 62 | 31
  Serious TEAEs | 31 | 12
  TEAEs >= Grade 3 | 48 | 17
  TEAEs Leading to Treatment Discontinuation | 18 | 6
  TEAEs Leading to Death Excluding Death Due to Disease Under Study | 3 | 0

9. Secondary Outcome: Serum Concentrations of Ociperlimab
Description: Serum samples were assayed for ociperlimab concentrations using a validated immunoassay. This outcome measure was not analyzed for Arm B as ociperlimab was not administered in Arm B.
Time Frame: Predose on Day 1 of Cycles 1, 2, 5, 9 and 17; Post dose on Day 1 of Cycles 1 and 5 and Safety Follow-up Visit (i.e., up to 30 days after last dose [up to 27 months]) (each cycle duration = 21-days)
Population: Analysis was performed on Pharmacokinetics (PK) analysis set that included all participants who received at least 1 dose of any component of study drugs as per the protocol, and for whom any post dose PK data was available. Here, "Overall number of participants analyzed" = participants with available data for this outcome measure and "number analyzed" signifies participants with available data for each specified category at respective visit.
Measure: Mean (Standard Deviation); unit: micrograms per milliliters (mcg/mL)
Arm/Group | Arm A: Ociperlimab + Tislelizumab + BAT1706
Number analyzed (Participants) | 61
micrograms per milliliters (mcg/mL)
  Cycle 1 Day 1: Pre-dose | 0.00 (0.000)
  Cycle 1 Day 1: Post-dose | 287.15 (50.203)
  Cycle 2 Day 1: Pre-dose: number analyzed (Participants) | 55
  Cycle 2 Day 1: Pre-dose | 39.82 (16.896)
  Cycle 5 Day 1: Pre-dose: number analyzed (Participants) | 44
  Cycle 5 Day 1: Pre-dose | 68.23 (28.422)
  Cycle 5 Day 1: Post-dose: number analyzed (Participants) | 46
  Cycle 5 Day 1: Post-dose | 385.22 (79.227)
  Cycle 9 Day 1: Pre-dose: number analyzed (Participants) | 29
  Cycle 9 Day 1: Pre-dose | 79.83 (30.614)
  Cycle 17 Day 1: Pre-dose: number analyzed (Participants) | 16
  Cycle 17 Day 1: Pre-dose | 78.16 (29.558)
  Safety Follow-up: Post Dose: number analyzed (Participants) | 15
  Safety Follow-up: Post Dose | 34.54 (28.961)

10. Secondary Outcome: Serum Concentrations of Tislelizumab
Description: Serum samples were assayed for tislelizumab concentrations using a validated immunoassay.
Time Frame: as for outcome 9
Population: Analysis was performed on PK analysis set. Here, "Overall number of participants analyzed" = participants with available data for this outcome measure and "number analyzed" signifies participants with available data for each specified category at respective visit.
Measure: Mean (Standard Deviation); unit: micrograms per milliliters (mcg/mL)
Arm/Group | Arm A: Ociperlimab + Tislelizumab + BAT1706 | Arm B: Tislelizumab + BAT1706
Number analyzed (Participants) | 61 | 30
micrograms per milliliters (mcg/mL)
  Cycle 1 Day 1: Pre-dose: number analyzed (Participants) | 59 | 30
  Cycle 1 Day 1: Pre-dose | 0.00 (0.000) | 0.00 (0.000)
  Cycle 1 Day 1: Post-dose | 69.63 (11.923) | 67.69 (12.545)
  Cycle 2 Day 1: Pre-dose: number analyzed (Participants) | 53 | 25
  Cycle 2 Day 1: Pre-dose | 19.65 (6.348) | 17.70 (5.875)
  Cycle 5 Day 1: Pre-dose: number analyzed (Participants) | 44 | 20
  Cycle 5 Day 1: Pre-dose | 38.14 (13.908) | 36.62 (11.920)
  Cycle 5 Day 1: Post-dose: number analyzed (Participants) | 46 | 19
  Cycle 5 Day 1: Post-dose | 106.93 (22.321) | 103.21 (21.305)
  Cycle 9 Day 1: Pre-dose: number analyzed (Participants) | 28 | 15
  Cycle 9 Day 1: Pre-dose | 43.82 (16.823) | 42.00 (16.495)
  Cycle 17 Day 1: Pre-dose: number analyzed (Participants) | 17 | 10
  Cycle 17 Day 1: Pre-dose | 39.35 (14.060) | 44.01 (21.788)
  Safety Follow-up: Post Dose: number analyzed (Participants) | 15 | 9
  Safety Follow-up: Post Dose | 23.90 (16.674) | 25.66 (26.011)

11. Secondary Outcome: Serum Concentrations of BAT1706
Description: Serum samples were assayed for BAT1706 concentrations using a validated immunoassay.
Time Frame: as for outcome 9
Population: Analysis was performed on PK analysis set. Here, "number analyzed" signifies participants with available data for each specified category at respective visit.
Measure: Mean (Standard Deviation); unit: micrograms per milliliters (mcg/mL)
Arm/Group | Arm A: Ociperlimab + Tislelizumab + BAT1706 | Arm B: Tislelizumab + BAT1706
Number analyzed (Participants) | 62 | 31
micrograms per milliliters (mcg/mL)
  Cycle 1 Day 1: Pre-dose: number analyzed (Participants) | 60 | 31
  Cycle 1 Day 1: Pre-dose | 0.00 (0.000) | 0.00 (0.000)
  Cycle 1 Day 1: Post-dose | 319.29 (58.599) | 321.03 (56.151)
  Cycle 2 Day 1: Pre-dose: number analyzed (Participants) | 54 | 24
  Cycle 2 Day 1: Pre-dose | 63.28 (19.302) | 55.30 (20.999)
  Cycle 5 Day 1: Pre-dose: number analyzed (Participants) | 43 | 18
  Cycle 5 Day 1: Pre-dose | 113.97 (37.045) | 112.79 (34.114)
  Cycle 5 Day 1: Post-dose: number analyzed (Participants) | 45 | 17
  Cycle 5 Day 1: Post-dose | 432.60 (86.670) | 410.71 (90.747)
  Cycle 9 Day 1: Pre-dose: number analyzed (Participants) | 22 | 14
  Cycle 9 Day 1: Pre-dose | 113.72 (38.039) | 120.55 (43.141)
  Cycle 17 Day 1: Pre-dose: number analyzed (Participants) | 15 | 10
  Cycle 17 Day 1: Pre-dose | 111.29 (31.055) | 123.36 (44.184)
  Safety Follow-up: Post Dose: number analyzed (Participants) | 25 | 17
  Safety Follow-up: Post Dose | 59.74 (40.020) | 81.42 (79.696)

12. Secondary Outcome: Number of Participants With Antidrug Antibodies (ADAs) to Ociperlimab, Tislelizumab, and BAT1706
Description: Serum samples were tested for the presence of ADAs to ociperlimab, tislelizumab and BAT1706 using a validated immunoassay. The analysis included: Treatment-emergent ADA: sum of treatment-boosted ADA patients and treatment-induced ADA participants as a percentage of the ADA-evaluable participants population; Treatment-boosted ADA: Baseline-positive ADA-evaluable patients with significant increases (4-fold or higher) in ADA titer after drug administration during the treatment or follow-up observation period; and Treatment-induced ADA: ADA-evaluable participants that were ADA-negative at baseline and ADA-positive after drug administration during the treatment or follow-up observation period.
Time Frame: Up to 27 months
Population: Analysis was performed on the Immunogenicity analysis set that included all participants who received at least 1 dose of any component of study drugs and for whom both baseline ADA and >=1 post-baseline ADA result was available. Here, "0" in the number analyzed field signifies that participants in Arm B were not assessed for anti-ociperlimab ADAs since they did not receive ociperlimab.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Ociperlimab + Tislelizumab + BAT1706 | Arm B: Tislelizumab + BAT1706
Number analyzed (Participants) | 57 | 29
Participants
  Treatment-emergent ADA: Ociperlimab: number analyzed (Participants) | 57 | 0
  Treatment-emergent ADA: Ociperlimab | 1 |
  Treatment boosted ADA: Ociperlimab: number analyzed (Participants) | 57 | 0
  Treatment boosted ADA: Ociperlimab | 0 |
  Treatment induced ADA: Ociperlimab: number analyzed (Participants) | 57 | 0
  Treatment induced ADA: Ociperlimab | 1 |
  Treatment-emergent ADA: Tislelizumab | 22 | 18
  Treatment boosted ADA: Tislelizumab | 1 | 2
  Treatment induced ADA: Tislelizumab | 21 | 16
  Treatment-emergent ADA: BAT1706 | 1 | 3
  Treatment boosted ADA: BAT1706 | 0 | 0
  Treatment induced ADA: BAT1706 | 1 | 3

ADVERSE EVENTS:
Time Frame: All cause-mortality data was collected from randomization through end of the study (i.e. up to 29 months). Serious adverse events (SAEs) and non-serious AEs (NSAEs) data were collected from the date of the first dose of study drug up to 30 days after last dose of study drug (up to 27 months)
Description: All-cause mortality data was analyzed for all randomized participants. SAEs, and NSAEs data analysis were performed on safety analysis set.
Arm/Group | Arm A: Ociperlimab + Tislelizumab + BAT1706 | Arm B: Tislelizumab + BAT1706
All-Cause Mortality (participants affected / at risk) | 28/62 | 14/32
Serious Adverse Events (participants affected / at risk) | 31/62 | 12/31
Other Adverse Events (participants affected / at risk) | 61/62 | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Ociperlimab + Tislelizumab + BAT1706 (N=62) | Arm B: Tislelizumab + BAT1706 (N=31)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial injury (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Haemobilia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1)
Biliary tract infection (Infections and infestations) | 2 (3) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Peritonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Blood creatine phosphokinase MB increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tumour rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Scrotal inflammation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Ociperlimab + Tislelizumab + BAT1706 (N=62) | Arm B: Tislelizumab + BAT1706 (N=31)
Anaemia (Blood and lymphatic system disorders) | 13 (20) | 4 (5)
Coagulopathy (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 2 (5) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (5) | 4 (4)
Angina pectoris (Cardiac disorders) | 2 (2) | 0 (0)
Bundle branch block right (Cardiac disorders) | 0 (0) | 1 (2)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial injury (Cardiac disorders) | 2 (3) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (2) | 0 (0)
Sinus arrhythmia (Cardiac disorders) | 0 (0) | 1 (2)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 1 (2) | 2 (6)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 7 (9) | 9 (9)
Thyroiditis subacute (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 3 (3) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Refraction disorder (Eye disorders) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1)
Ascites (Gastrointestinal disorders) | 6 (6) | 3 (4)
Constipation (Gastrointestinal disorders) | 7 (9) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 10 (12) | 10 (13)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (2)
Gingival bleeding (Gastrointestinal disorders) | 2 (2) | 3 (4)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 0 (0) | 1 (1)
Loose tooth (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Oral discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 3 (4) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (5) | 2 (2)
Asthenia (General disorders) | 4 (4) | 1 (2)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 8 (11) | 3 (3)
Malaise (General disorders) | 3 (3) | 2 (2)
Oedema peripheral (General disorders) | 6 (6) | 5 (5)
Pain (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 13 (26) | 4 (6)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatitis cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (2)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (2) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 1 (2)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
COVID-19 (Infections and infestations) | 12 (34) | 6 (6)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (3) | 2 (2)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 0 (0) | 2 (4)
Pharyngitis (Infections and infestations) | 3 (3) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 1 (2)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 3 (3)
Urinary tract infection (Infections and infestations) | 4 (5) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 23 (40) | 8 (15)
Androgens abnormal (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 26 (49) | 9 (13)
Bile acids increased (Investigations) | 0 (0) | 1 (2)
Bilirubin conjugated increased (Investigations) | 1 (1) | 2 (2)
Bilirubin urine present (Investigations) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 10 (17) | 1 (1)
Blood bilirubin increased (Investigations) | 10 (17) | 8 (12)
Blood corticotrophin increased (Investigations) | 0 (0) | 1 (1)
Blood creatine phosphokinase MB increased (Investigations) | 2 (2) | 2 (3)
Blood creatine phosphokinase increased (Investigations) | 7 (16) | 2 (5)
Blood creatinine increased (Investigations) | 5 (5) | 1 (1)
Blood fibrinogen increased (Investigations) | 3 (4) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 6 (17) | 2 (2)
Blood pressure increased (Investigations) | 2 (3) | 1 (2)
Blood thyroid stimulating hormone increased (Investigations) | 2 (2) | 0 (0)
Blood urea increased (Investigations) | 2 (2) | 0 (0)
Cortisol decreased (Investigations) | 3 (3) | 0 (0)
Cortisol increased (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 7 (9) | 2 (2)
Glomerular filtration rate decreased (Investigations) | 1 (2) | 1 (1)
Glucose urine present (Investigations) | 2 (2) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (2) | 0 (0)
Myocardial necrosis marker increased (Investigations) | 2 (2) | 1 (1)
Neutrophil count decreased (Investigations) | 4 (6) | 2 (3)
Neutrophil count increased (Investigations) | 2 (3) | 0 (0)
Platelet count decreased (Investigations) | 23 (59) | 8 (15)
Platelet count increased (Investigations) | 2 (2) | 0 (0)
Protein urine present (Investigations) | 2 (5) | 1 (1)
Prothrombin time prolonged (Investigations) | 1 (1) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 3 (3)
Troponin I increased (Investigations) | 0 (0) | 1 (1)
Troponin T increased (Investigations) | 1 (1) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 1 (1)
Urinary occult blood positive (Investigations) | 0 (0) | 1 (1)
Urobilinogen urine increased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 8 (8) | 4 (4)
Weight increased (Investigations) | 2 (5) | 2 (2)
White blood cell count decreased (Investigations) | 9 (17) | 3 (4)
White blood cell count increased (Investigations) | 3 (4) | 1 (1)
White blood cells urine positive (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 9 (11) | 5 (5)
Electrolyte imbalance (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 (5) | 2 (4)
Hyperuricaemia (Metabolism and nutrition disorders) | 11 (22) | 2 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 12 (17) | 10 (16)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (6) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 10 (13) | 4 (8)
Hyponatraemia (Metabolism and nutrition disorders) | 8 (8) | 3 (7)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 7 (8) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Lacunar infarction (Nervous system disorders) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (6) | 3 (4)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (3) | 3 (3)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 1 (1)
Proteinuria (Renal and urinary disorders) | 24 (36) | 16 (29)
Renal impairment (Renal and urinary disorders) | 0 (0) | 2 (2)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Pruritus genital (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 3 (5) | 0 (0)
Immune-mediated dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Leukoderma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (15) | 2 (2)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 15 (17) | 6 (7)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 23 (34) | 15 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2021-03-03): https://cdn.clinicaltrials.gov/large-docs/97/NCT04948697/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/97/NCT04948697/SAP_001.pdf